CLINICAL TRIAL: NCT02640586
Title: Predicting Neoadjuvant Therapy Response of Rectal Cancer With MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Ying-Shi (Other)
Responsible Party: Sponsor-Investigator, Sun Ying-Shi, Chairman of Department of Radiology, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PNTRRC-MRI
Record Dates: First submitted 2015-12-17; First posted 2015-12-29 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessing response with MRI (Experimental): Preoperative chemo-radiotherapy as standard treatment. Neoadjuvant therapy (long course intensity modulated radio-chemotherapy, GTV 50.6Gy, totally 22 fractions; Capecitabine 825mg/m2 /bid by oral administration).
  Three MR examinations: first MRI taken within 1 week before preoperative chemo-radiotherapy; second MRI taken between 14-16days after the initiation of radio-chemotherapy; third MRI taken 7-9 weeks after the completion of preoperative chemo-radiotherapy.
  All patients are scheduled to receive total mesorectal excision surgery 12-14 weeks after the completion of preoperative chemo-radiotherapy.
  Interventions: Device: three MR examination

INTERVENTIONS:
Device: three MR examination — Three MR examinations: first MRI taken within 1 week before preoperative chemo-radiotherapy; second MRI taken between 14-16days after the initiation of radio-chemotherapy; third MRI taken 7-9 weeks after the completion of preoperative chemo-radiotherapy.
  Other Names: imaging

SUMMARY:
The purpose of this study is to investigate if MRI scans performed after neoadjuvant radiotherapy can predict the therapeutic response of rectal cancer following preoperative chemo-radiotherapy. This will help doctors to better tailor treatments for rectal cancer in the future.

DETAILED DESCRIPTION:
We proposed to constructed multi-parameter predictive model for predicting therapeutic response and pathological complete response(pCR) of patients with rectal cancer who received neoadjuvant chemoradiation. MR radiomics,convolutional neural networks, morphological parameters and quantitative functional parameters derived from diffusion-weighted MR images will be integrated for model construction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* T3/4 or node positive biopsy-proved primary rectal cancer
* Suitable for pre-operative chemoradiotherapy and surgical resection
* No contraindication to MRI
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History or concurrent of other cancer
* Previous therapy to pelvis
* Unable/unwilling to have MRI
* Pacemaker or implanted defibrillator
* Pregnancy, lactation or inadequate contraception
* Patients with a history of psychological illness or condition such as to interfere with the patient's ability to understand requirements of the study
* Unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1614 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of eary MRI (14-16 days MRI) for assessing pathological complete response(pCR) at surgery | 2 years
  A scoring system for predicting pCR will be developed based on MRI parameters and their changes between baseline and early MRI. No viable cancer cells seen in the resection specimen is regarded as pCR
Predictive value of preoperative MRI(7-9 weeks after the completion of preoperative chemo-radiotherapy) for assessing pCR | 2 years
  A scoring system for predicting pCR will be developed based on MRI parameters

SECONDARY OUTCOMES:
Predictive value of eary MRI (14-16 days after initiation of preoperative radio-chemotherapy) for assessing pathological response according to Tumour Regression Grade (TRG) | 2 years
  A scoring system for predicting pathological response will be developed based on MRI parameters and their changes between baseline and early MRI.TRG1 is regarded as responder, and TRG2/3 is regarded as non-responder.
Feasibility of conducting MRI scans at 7-9 weeks after preoperative radio-chemotherapy | 2 years
  This will be assessed in terms of whether MR imaging at 7-9 weeks after preoperative radio-chemotherapy adds any additional predictive value to imaging performed 14-16 days after initiation of preoperative radio-chemotherapy.
MRI-predicted pCR and MRI-predicted response on long-term disease control and survival | 3 years
  3 years disease-free survival and overall survival will be assessed
Predictive value of preoperative MRI(7-9 weeks after the completion of preoperative chemo-radiotherapy) for assessing pathological response according to Tumour Regression Grade (TRG) | 2 years
  A scoring system for predicting pathological response will be developed based on MRI parameters and their changes between baseline and early MRI.TRG1 is regarded as responder, and TRG2/3 is regarded as non-responder.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Shi Sun, MD, Study Chair — No.52 Fu Cheng Road, Hai Dian District, Beijing, 10142
Locations (11):
- China (11):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Capital Medical University, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences, Cancer Hospital & Institute, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangxi Cancer Hospital, Guilin, Guangxi
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Shanxi Cancer Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No